CLINICAL TRIAL: NCT03162471
Title: Impact of Preoperative Astigmatism on Corneal Biomechanics and Accurate Intraocular Pressure Measurement After Micro-incision Phacoemulsification
Brief Title: How Astigmatism Influences Corneal Biomechanics and Intraocular Pressure
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Zofia Pniakowska, M.D., Medical University of Lodz
Other Study IDs: RNN/166/17/KE
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Corneal Astigmatism; Intraocular Pressure; Cataract Senile
Keywords: Corneal astigmatism; Cataract surgery; Corneal hysteresis; Corneal resistance factor; Intraocular pressure
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: non-contact measurement of intraocular pressure — Non-contact measurement of corneal biomechanical properties and intraocular pressure with an Ocular Response Analyzer. Parameters measured: corneal hysteresis (CH), corneal resistance factor (CRF), Goldman-correlated IOP (IOPg), corneal compensated IOP (IOPcc) and waveform score (WS).

SUMMARY:
The aim of the study was to identify whether preoperative corneal astigmatism can influence corneal biomechanics and the assessment of intraocular pressure (IOP) following micro-incision phacoemulsification.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis and qualification for cataract surgery, corneal astigmatism of equal to or less than 2.25 Dcyl

Exclusion Criteria:

* corneal astigmatism higher than 2.25 Dcyl, history of any other corneal disease (infection, trauma, ulceration, autoimmune inflammation, Fuchs Dystrophy, keratoconus, corneal scars, preoperative insufficiency of corneal endothelium), glaucoma and chronic use of non-glaucoma eye drops, blepharitis, dry eye, use of contact lenses diabetes or a history of corneal refractive surgery

Ages: 52 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 39 patients diagnosed with cataracts were enrolled in the study
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
change of corneal compensated IOP (IOPcc) | Parameter measured preoperatively and one day, one week, one month postoperatively
  Intraocular pressure and corneal biomechanical properties were measured using an Ocular Response Analyzer.

SECONDARY OUTCOMES:
change of corneal hysteresis (CH) | Parameter measured preoperatively and one day, one week, one month postoperatively
  Intraocular pressure and corneal biomechanical properties were measured using an Ocular Response Analyzer.
change of corneal resistance factor (CRF) | Parameter measured preoperatively and one day, one week, one month postoperatively
  Intraocular pressure and corneal biomechanical properties were measured using an Ocular Response Analyzer.
change of Goldman-correlated IOP (IOPg) | Parameter measured preoperatively and one day, one week, one month postoperatively
  Intraocular pressure and corneal biomechanical properties were measured using an Ocular Response Analyzer.
change of waveform score (WS) | Parameter measured preoperatively and one day, one week, one month postoperatively
  Intraocular pressure and corneal biomechanical properties were measured using an Ocular Response Analyzer.

IPD SHARING:
Plan to Share IPD: No